CLINICAL TRIAL: NCT04604886
Title: The Consistency of Cardiac Output Measured by Pulmonary Artery Catheter and LiDCO in Cardiac Surgical Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: COMPACT-LiDCO
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Cardiac Surgery; Cardiac Output
Keywords: Hemodynamic Monitoring; Pulmonary artery catherization; LiDCO

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive Leg Raising (Experimental): Passive leg raising (PLR) test is used to predict fluid responsiveness, which is performed by raising the legs of the patient to 45°. Cardiac output will be collected from both PAC and LiDCO before and after PLR.
  Interventions: Diagnostic Test: Passive Leg Raising
- Dobutamine stress test (Experimental): Dobutamine is a selective beta 1 receptor agonist. It [<10 ug/(kg.min)] can effectively increase myocardial contractility.
  Interventions: Diagnostic Test: Dobutamine stress test

INTERVENTIONS:
Diagnostic Test: Passive Leg Raising — Passive leg raising is induced by rasing the legs of patients to 45° from horizontal position.
  Arms: Passive Leg Raising
Diagnostic Test: Dobutamine stress test — Dobutamine was infused intravenously at the initial dose of 2.5 ug/kg/min. hemodynamic data were recorded from PAC and LiDCO after 5-10 minutes of continuous infusion.
  Arms: Dobutamine stress test

SUMMARY:
1. To evaluate the consistency of cardiac output measured by pulmonary artery catheter and LiDCO in cardiac surgical patients
2. To evaluate whether different hemodynamic monitoring methods can accurately detect the trend of cardiac output changes

DETAILED DESCRIPTION:
Close monitoring of cardiac output (CO), especially in patients before and after intervention(such as volume expansion, diuresis, vasoconstriction, vasodilation therapy), could help to adjust the treatment strategy in cardiac surgical patients. Pulmonary artery catherization (PAC) has been used for hemodynamic monitoring for more than four decades. In spite of its invasiveness, it remains the clinical reference method for the assessment of CO at the bedside. Nowadays, many less invasive alternatives, such as LiDCO Rapid Pulse Contour Analysis System (LiDCO Ltd., Cambridge, United Kingdom), are already available on market. However, consistency between different hemodynamic monitoring results still raise concern. And whether hemodynamic monitoring could accurately detect the changes of these parameters before and after intervention is an important issue in clinical practice. In this study, the investigators are going to collect CO and changes of CO from PAC and LiDCO before and after intervention (passive leg raising and dobutamine stress test) in cardiac surgical patients. Our resulst could provide important reference for cardiac surgical patients how to choose appropriate hemodynamic monitoring tools and how to interpret the results of hemodynamic monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. cardiac surgery
2. hemodynamic monitoring (PAC, LiDCO)
3. mechanical ventilation

Exclusion Criteria:

1. cardiac arrhythmia
2. moderate to severe aortic, mitral and tricuspid regurgitation
3. IABP
4. ECMO

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Baseline Cardiac Output measurement | within1 minute at baseline position
  Cardiac Output measured at baseline position (horizontal position)
Cardiac Output measurement after PLR | 1 minute after PLR
  Cardiac Output measured after PLR
Cardiac Output measurement after Dobutamine stress test | 5 minutes after dobutamine stress test
  Cardiac Output measured after dobutamine stress test

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Luo, Doctor, Study Chair — Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, China